CLINICAL TRIAL: NCT05132140
Title: Peripheral Choroidal Response to Pure Defocus and Oriented Blur Conditions
Brief Title: Peripheral Choroidal Layer Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Geunyoung Yoon, Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00003210
Record Dates: First submitted 2021-11-11; First posted 2021-11-24 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- normal healthy group (Experimental): Adaptive optics system: this system controls the optical quality of the eye at the peripheral visual field temporarily.
  Interventions: Device: adaptive optics system

INTERVENTIONS:
Device: adaptive optics system — the system consists of a wavefront sensor and a deformable mirror that measure and correct (or modify) the eye's optical imperfections (aberrations).

SUMMARY:
The study aims to examine how the vascular layer of the eyeball (choroidal layer) responds when part of the visual field is exposed to specially generated visual stimulus. The study goal will be accomplished by producing specific blur visual stimulus at a particular visual field position and measure any consistent thickness change pattern in the choroidal layer.

We propose to test the hypothesis that regional changes in the choroidal thickness may be induced differently after short-term exposure to specific visual stimuli.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is between the ages of 18 and 40 yrs old
* Has normal best corrected visual acuity being 20/20 or better
* Has spherical refractive error between +1.00D and -6.00D.
* Is capable of fixating on the target.
* Has no prior ocular surgery.
* Has no ocular pathology except keratoconus.
* Can tolerate dilating eye drops

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Does not fall within above mentioned age group.
* Has chronic or systemic eye disease that would interfere with pupil dilation via eye drops.
* Underwent ocular surgeries or history of ocular trauma
* Has shallow anterior chamber angle and/or glaucoma.
* Has clinically significant dry eye.
* Has signs of any choroidal or retinal pathology, and abnormalities in the visual pathway
* Has spherical refractive error that exceeds the limits outlined above.
* Has binocular anomalies (e.g. convergence insufficiency, strabismus, pseudo-myopia, amblyopia).
* Is an adult unable to consent
* Is an individual who is not yet adult (infants, children, teenagers)
* Is a pregnant woman
* Is a prisoner
* Is a student for whom you have direct access to/influence on grades
* Is an economically and/or educationally disadvantaged person

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
choroidal thickness | up to 60 mins
  A commercially available optical coherence tomography system will be used to measure changes in choroidal layer thickness before and after manipulating the peripheral optics.

CONTACTS AND LOCATIONS:
Overall Officials: Geunyoung Yoon, PhD, Principal Investigator — University of Houston

IPD SHARING:
Plan to Share IPD: No